CLINICAL TRIAL: NCT00270777
Title: Low Dose Adrenaline, Promethazine, & Hydrocortisone (Alone and in Combination) to Prevent Acute Adverse Reactions to Antivenom in People Bitten by Snakes: Randomised, Double Blind, Placebo-Controlled Trial
Brief Title: Improving Safety of Antivenom in People Bitten by Snakes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kelaniya (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 178A07
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Snake Bites
Keywords: Controlled trial; Snake bite; Safety; Antivenom
MeSH Terms: conditions — Snake Bites | interventions — Epinephrine; Promethazine; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: adrenaline, promethazine, hydrocortisone

SUMMARY:
A study to increase the safety of polyvalent antivenom involving 1000 patients in three centres: low dose adrenaline, promethazine, & hydrocortisone (alone and in combination) to prevent acute adverse reactions to antivenom in people bitten by snakes: randomised, double blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Above 12 years of age
* Patients admitted to hospital after snake bite in whom antivenom is indicated
* Patients who give informed consent

Exclusion Criteria:

* Patients who are pregnant or nursing
* Patients who are currently taking beta- or alpha-adrenoceptor antagonists, or tricyclic antidepressants
* Patients in whom adrenaline may be contraindicated (this may include patients with the following: history of ischaemic heart disease, stroke, uncontrolled hypertension, and tachyarrhythmias)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Frequency of severe reactions to antivenom in the first 48 hours

SECONDARY OUTCOMES:
Frequency of moderate & severe reactions to antivenom in the first 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Asita de Silva, Principal Investigator — University of Kelaniya
Locations (1):
- Clinical Trials Unit, University of Kelaniya, Ragama, Sri Lanka

REFERENCES:
- [Derived] de Silva HA, Pathmeswaran A, Ranasinha CD, Jayamanne S, Samarakoon SB, Hittharage A, Kalupahana R, Ratnatilaka GA, Uluwatthage W, Aronson JK, Armitage JM, Lalloo DG, de Silva HJ. Low-dose adrenaline, promethazine, and hydrocortisone in the prevention of acute adverse reactions to antivenom following snakebite: a randomised, double-blind, placebo-controlled trial. PLoS Med. 2011 May;8(5):e1000435. doi: 10.1371/journal.pmed.1000435. Epub 2011 May 10. PMID 21572992